CLINICAL TRIAL: NCT02451410
Title: Impact of an Intervention to Improve Nutrition and Physical Activity in Preschoolers in Cuenca, Ecuador
Brief Title: An Intervention to Improve Nutrition and Physical Activity in Preschoolers in Cuenca, Ecuador
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Cuenca (Other)
Collaborators: Universidad de Antioquia (Other)
Responsible Party: Principal Investigator, Victoria Abril, Researcher, Universidad de Cuenca
Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: Intervention1
Record Dates: First submitted 2015-05-11; First posted 2015-05-22 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Obesity; Overweight; Underweight
Keywords: Nutrition; Physical activity; Overweight; Obesity; Malnutrition
MeSH Terms: conditions — Obesity; Overweight; Thinness; Motor Activity; Malnutrition | interventions — Nutritional Status; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nutrition and physical activity (Experimental): This arm includes all preschool classes receiving the educational and behavioral intervention to improve nutrition and physical activity
  Interventions: Other: Nutrition and physical activity

INTERVENTIONS:
Other: Nutrition and physical activity — The investigators will design an educational and behavioral program focused on health promotion. Didactic material will be developed for teachers and educational material will be developed for parents. For children, the investigators will design educational and playtime materials that encourage healthy eating and physical activity.

SUMMARY:
The aim of this study is to design and evaluate an educational and behavioral intervention focused on improving nutrition and physical activity habits among preschoolers in Cuenca, Ecuador, with the overarching goal of preventing overweight/obesity and promoting the formation of healthy nutrition/physical activity habits.

DETAILED DESCRIPTION:
In Ecuador and in the city of Cuenca, the prevalence of obesity is high (approximately 22% of the population). Simultaneously, there is high prevalence of chronic malnutrition (e.g., stunting). In a previous study in school-aged children in Cuenca, the prevalence of overweight or obese was 30%.

The objective of this study is to design an intervention to improve nutrition and physical activity habits and behaviors in preschoolers. The study will begin with a baseline survey that will be used to develop the educational and behavioral intervention. The intervention will consist of didactic material for teachers, educational material for parents, and activities for the children. The investigators will carry out the intervention over the course of the school year. The intervention will be primarily delivered in the preschool setting, but will also include workshops for parents.

The investigators hope that this study will help promote the health of children in Cuenca and can be a pilot study to test similar interventions in larger populations in Ecuador.

ELIGIBILITY:
Inclusion Criteria:

Any child attending a preschool of the municipality

Exclusion Criteria:

Any child whose parents decline inclusion in the study

Ages: 3 Years to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 307 (Actual)
Dates: Start 2015-09; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Fruit and vegetable consumption habits | Changes over 1 year (with 30-day recall). Assessment pre/post intervention (approx 9 months in between).
  Changes assessed using a pre-/post-intervention questionnaire evaluating the number of days per week fruits/vegetables were consumed as snacks at home.
Drinking habits | Changes over 1 year (with 30-day recall). Assessment pre/post intervention (approx 9 months in between).
  Changes assessed using a pre-/post-intervention questionnaire evaluating the number of days per week water, fruit juices, and soft drinks are consumed at home.
Screen time habits | Changes over 1 year (with 30-day recall). Assessment pre/post intervention (approx 9 months in between).
  Changes assessed using a pre-/post-intervention questionnaire evaluating weekly hours of time spent watching television, using the computer, and playing videogames at home.

SECONDARY OUTCOMES:
Nutritional status | 1 year. Assessment pre/post intervention (approx 9 months in between).
  Changes assessed using anthropometry

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Abril, PhD, Principal Investigator — Universidad de Cuenca
Locations (9):
- Ecuador (9):
  - Centro Infantil 12 de Abril, Cuenca
  - Centro Infantil 27 de Febrero, Cuenca
  - Centro Infantil 9 de Octubre, Cuenca
  - Centro Infantil El Arenal, Cuenca
  - Centro Infantil El Cebollar, Cuenca
  - Centro Infantil El Condor, Cuenca
  - Centro Infantil San Blas, Cuenca
  - Centro Infantil Sol de Talentos, Cuenca
  - Centro Infantil Totoracocha, Cuenca

REFERENCES:
- [Background] Abril V, Manuel-y-keenoy B, Sola R, Garcia JL, Nessier C, Rojas R, Donoso S, Arija V. Prevalence of overweight and obesity among 6-to 9-year-old school children in Cuenca, Ecuador: relationship with physical activity, poverty, and eating habits. Food Nutr Bull. 2013 Dec;34(4):388-401. doi: 10.1177/156482651303400404. PMID 24605689